CLINICAL TRIAL: NCT04974827
Title: A Single-arm, Multi-center Phase II Clinical Study of Camrelizumab Combined With Concurrent Chemoradiation in Patients With Cervical Cancer Who Had Recurrence of the Pelvic Wall After Surgery ± Abdominal Aortic Lymph Node Metastasis
Brief Title: A Study of Camrelizumab Combined With Concurrent Chemoradiation in Patients With Cervical Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hunan Cancer Hospital (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HNCHIIT003
Record Dates: First submitted 2021-07-05; First posted 2021-07-23 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-07

CONDITIONS: Cervical Cancer
Keywords: immunotherapy; PD-1 checkpoint inhibitor; concurrent chemoradiation
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — camrelizumab; Cisplatin; Carboplatin

STUDY DESIGN:
Intervention Model Description: Patients fulfilling Eligibility Criteria will be included in this study.Participants will be given intravenous administration of Camrelizumab (200mg) ,Cisplatin(40mg/m²) or Carboplatin(AUC 2) and Radiotherapy. After completing 5 cycles of concurrent chemoradiation, the Participants will continue to use camrelizumab as maintenance therapy until one year.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camrelizumab , Cisplatin or Carboplatin (Experimental): Participants will be given intravenous administration of Camrelizumab (200mg) ,Cisplatin(40mg/m²) or Carboplatin(AUC 2) and Radiotherapy. After completing 5 cycles of concurrent chemoradiation, the Participants will continue to use camrelizumab as maintenance therapy until one year.
  Interventions: Drug: Camrelizumab; Drug: Cisplatin or Carboplatin

INTERVENTIONS:
Drug: Camrelizumab — 200mg/3weeks
Drug: Cisplatin or Carboplatin — Cisplatin (40mg/m²), every week Carboplatin(AUC 2)

SUMMARY:
In this single-arm study, patient with cervical cancer who had recurrence of the pelvic wall after surgery ± Abdominal aortic lymph node metastasis will be included to evaluate the efficacy and safety of camrelizumab combined with concurrent chemoradiation and subsequent maintenance therapy

DETAILED DESCRIPTION:
The patient received neoadjuvant therapy once every three weeks for a total of seventeen cycles. From the first day of treatment, the patient will undergo concurrent chemoradiation for 5 weeks.The chemotherapy drug is cisplatin or carboplatin every week for 5 weeks. After the end of concurrent chemoradiation, the patient will continue to use camrelizumab as maintenance therapy until one year.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old
2. Understand the research procedures and content, and voluntarily sign informed consent
3. Cervical squamous cell carcinoma, adenocarcinoma or adenosquamous carcinoma confirmed by histology or cytology
4. Patients diagnosed as recurrent cervical cancer on the pelvic wall by histology or cytology. If histology or cytology is not available, provide clinical diagnosis in combination with medical history, laboratory examinations and imaging examinations (such as CT, MRI, PET/CT)
5. According to the RECIST 1.1 standard, the subject must have at least one measurable target lesion on the pelvic wall by CT or MRI (the longest diameter ≥10mm lesion, or the short diameter ≥15mm lymph node)
6. CT or MRI examination or PET-CT examination showed no distant metastasis
7. Expected survival period ≥ 3 months
8. ECOG score: 0-1
9. Participants need to provide sufficient formalin-fixed paraffin-embedded (FFPE) specimens or sections prepared from tumor archive tissues or fresh tissues that meet the testing standards, and are willing to perform tumor tissue biopsy when needed for PD-L1 Detection. The archived tissue must be a representative tumor specimen within three years, or an unstained serial section (not less than 4 pieces) of newly cut FFPE tumor tissue within six months, and relevant pathological reports of the above specimens must be provided. The methods of obtaining fresh tissue specimens can be surgical resection and biopsy. The methods of biopsy include but are not limited to core needle biopsy, endoscopic resection or clamp biopsy (enough tumor cells must be guaranteed> 100); Fine needle aspiration and liquid-based cytology (TCT) samples are not accepted (it means that there isn't a complete tissue structure and Participants only provide cell suspension and/or cell smears); Decalcified bone metastasis tumor tissue specimens are not accepted. For patients who are PD-L1 negative in the initial archived tumor tissue samples, after obtaining the patient's consent, a biopsy can be performed during screening to provide wax blocks or sections prepared from fresh tissues to retest PD-L1 status
10. The investigator assesses suitability for concurrent chemoradiation
11. The values of laboratory tests performed during the screening period must meet the following criteria Hemoglobin (HGB) ≥90g/L Absolute neutrophil count (ANC) ≥1.5×109/L Platelet (PLT) ≥100×109/L Total bilirubin (TBIL)≤1.5×ULN (Gilbert syndrome allows ≤5×ULN) Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5×ULN Serum creatinine (Cr) ≤ 1.5 × ULN or endogenous creatinine clearance ≥ 50mL/min
12. Thyroid function index: free thyroxine (FT3/FT4) in the normal range
13. Subjects can be followed up on schedule, can communicate well with the investigator and can complete the study in accordance with the regulations of this study

Exclusion Criteria:

1. Histological examination results are small cell (neuroendocrine) cervical cancer and mucinous adenocarcinoma
2. CT, MRI or PET-CT examination shows diffuse pelvic metastasis
3. CT, MRI or PET-CT examination shows distant metastasis (excluding retroperitoneal lymph node metastasis)
4. Simple vaginal recurrence
5. Active central nervous system (CNS) metastases, including symptomatic brain metastases,meningeal metastases or spinal cord compression, etc.Asymptomatic brain metastases can be included in the group (no progression for at least 4 weeks after radiotherapy and/or no neurological symptoms or signs after surgical resection, no need for treatment with glucocorticoids, anticonvulsants or mannitol)
6. Systemic chemotherapy, targeted therapy, anti-tumor biological therapy (such as tumor vaccine, cytokine or growth factor, etc.) have been performed before the study drug
7. The effect of major surgery or severe trauma before study medication has been eliminated within 14 days(Those who have undergone local anesthesia or percutaneous needle biopsy within 7 days and have recovered can be included in the group)
8. Participants received systemic corticosteroids (prednisone>10mg/day or equivalent dose) or other immunosuppressive drugs within 14 days before the study medication
9. A history of active and known autoimmune diseases, including but not limited to systemic lupus erythematosus, psoriasis, rheumatoid arthritis, inflammatory bowel disease, Hashimoto's thyroiditis, etc. Except for type I diabetes, hypothyroidism that can be controlled only by hormone replacement therapy, skin diseases that do not require systemic treatment (such as vitiligo), and controlled celiac disease
10. Complications that need to be treated with immunosuppressive drugs, or Complications that need to be treated systemically with an immunosuppressive dose (prednisone> 10 mg/day or equivalent dose of similar drugs). In the absence of active autoimmune diseases, inhaled or topical steroids and doses> 10mg/day of prednisone or equivalent doses of similar drugs are allowed
11. Uncontrolled hypertension (systolic blood pressure> 140 mmHg and/or diastolic blood pressure> 90 mmHg) or pulmonary hypertension or unstable angina pectoris; myocardial infarction or bypass or stent surgery within 6 months before administration. A history of chronic heart failure that meets NYHA standards 3-4; clinically significant valvular disease; Severe arrhythmia requiring treatment, including QTc interval ≥470ms (calculated by Fridericia formula); left ventricular ejection fraction (LVEF) <50%;Cerebrovascular accident (CVA) or transient ischemic attack (TIA) within 6 months before administration.
12. Combined with other serious medical diseases, including but not limited to uncontrolled diabetes, active peptic ulcer, active bleeding, etc.
13. Patients with active infection who need systemic treatment
14. Patients with previous or current active tuberculosis infection
15. The patient has a history of interstitial lung disease
16. Symptomatic and uncontrollable serous effusion such as peritoneal effusion, pleural effusion or pericardial effusion
17. Human immunodeficiency virus antibody (HIV-Ab) positive; patients with active syphilis infection; hepatitis C antibody (HCV-Ab) positive, and hepatitis C virus RNA quantification> the upper limit of normal value of detection unit; hepatitis B virus surface antigen (HBsAg) is positive, and hepatitis B Virus detection value> upper limit of normal value of detection unit
18. Adverse reactions caused by previous treatment have not recovered to grade 1 or below (CTCAE5.0) (except for hair loss and grade 2 neurotoxicity caused by chemotherapy drugs)
19. Previously treated with anti-PD-1 antibody, anti-PD-L1 antibody, anti-PD-L2 antibody or anti-CTLA-4 antibody (or any other antibody that acts on T cell co-stimulation or checkpoint pathway)
20. Radiotherapy has been performed on the area to be irradiated in the past
21. Have used live vaccines or attenuated vaccines within 28 days before study medication
22. Participants have used other investigational drug treatments or investigational devices within 30 days before the study medication
23. People with a history of drug abuse or drug abuse
24. Have a clear history of neurological or mental disorders, such as epilepsy, dementia, and poor compliance
25. Women who are breastfeeding and do not agree to stop breastfeeding
26. Patients are known to be allergic to recombinant humanized PD-1 monoclonal antibody or any of its excipients; patients are known to have a history of allergic diseases or have severe allergies
27. The investigator believes that the patient is not suitable for participating in this clinical research for various other reasons

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2021-05-20 (Actual); Primary Completion 2023-05-20 (Estimated); Study Completion 2023-05-20 (Estimated)

PRIMARY OUTCOMES:
Complete remission rate (CR) | immediately after the concurrent chemoradiation
  Evaluate the efficacy of camrelizumab combined with Concurrent chemoradiation in patients with cervical cancer who had recurrence of the pelvic wall after surgery ± Abdominal aortic lymph node metastasis. Use RECIST 1.1 evaluation criteria for evaluation and the unit is '%'.

SECONDARY OUTCOMES:
objective response rate (ORR) duration of response in CR patients (DOR) disease control rate (DCR) progression-free survival (PFS) overall survival (OS) other efficacy indicators | immediately after the concurrent chemoradiation
  The proportion of patients whose tumor volume has shrunk to a predetermined value and can maintain the minimum time limit is the sum of the proportions of complete remission and partial remission. Use RECIST 1.1 evaluation criteria for evaluation and the unit is '%'.
Disease Control Rate (DCR) | 1 year
  The proportion of patients whose tumors have shrunk or stabilized for a certain period of time, including complete remission, partial remission and stable cases. Use RECIST 1.1 evaluation criteria for evaluation and the unit is '%'.
overall survival (OS) | 1 year
  Time from receiving treatment to death (for any reason). Evaluation based on follow-up and the unit is 'years'.
duration of response (DOR) | 1 year
  It refers to the time from the first evaluation of the tumor as CR or PR to the first evaluation as PD (Progressive Disease) or death from any cause. Use RECIST 1.1 evaluation criteria for evaluation and the unit is 'years'.
Progression-free survival (PFS) | 1 year
  The time span from the beginning of treatment of the tumor to the appearance of secondary growth of the tumor. It means that the tumor has basically not progressed at this stage. Use RECIST 1.1 evaluation criteria for evaluation and the unit is 'years'.

CONTACTS AND LOCATIONS:
Overall Officials: Chaoxia c Liu, Principal Investigator — Hunan Cancer Hospital
Locations (1):
- Hunan cancer Hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research
Supporting Information: Study Protocol
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: please contact the principal investigator of this study or correspondence author of published work